CLINICAL TRIAL: NCT04169425
Title: Laparoscopic Surgery of Rectal Cancer and Ileostomy. Technological Progress in Relation to New Minimally Invasive Treatment Methods and the Incidence of Complications.
Brief Title: Laparoscopic Surgery of Rectal Cancer and Ileostomy
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Vincenzo La Vaccara, Principal Investigator, Campus Bio-Medico University
Other Study IDs: 11.17 OSS Comet CBM
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Ileostomy - Stoma; Ileostomy; Complications; Leakage, Anastomotic
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients who underwent to laparoscopic TME, with elective diverting ileostomy for rectal cancer
  Interventions: Procedure: elective diverting ileostomy
- Group 2: patients who underwent to laparoscopic TME, without elective diverting ileostomy for rectal cancer

INTERVENTIONS:
Procedure: elective diverting ileostomy
  Groups: Group 1

SUMMARY:
Elective diverting ileostomy may reduce consequences of anastomotic failure in laparoscopic TME. Aiming to evaluate the effectiveness of elective diverting ileostomy, its impact on the incidence and clinical behavior of anastomotic leakage and the complications related to its presence and take down were analyzed.

DETAILED DESCRIPTION:
From a prospective collected database, data regarding patients who underwent to laparoscopic TME, with (Group 1) or without (Group 2) elective diverting ileostomy for rectal cancer from 2012 to 2017 at University Campus Bio-Medico di Roma, have been retrospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years and over)
* patients submitted to elective Anterior Rectal Resection

Exclusion Criteria:

* chronic use of immunosuppressant agents
* urgent surgery

Ages: 67 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who underwent to laparoscopic TME, for rectal cancer from 2012 to 2017 at University Campus Bio-Medico di Roma.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-01-02; Primary Completion 2017-12-22 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with anastomotic leakage | 90 days
  Leakage was defined on the basis of perianastomotic drain appearance and/or of radiological findings during postoperative X-Ray or abdominal CT scan enema

SECONDARY OUTCOMES:
Number of participants with post-operative complications | 90 days
  post-operative complication in patients submitted to Anterior Rectal Resection
Number of participants with fever Surgical site infection Abdominal collections Anastomotic leakage Anastomotic bleeding Perforation Anastomotic stenosis Number of participants with fever | 90 days
  post-operative fever in patients submitted to Anterior Rectal Resection
Number of participants with surgical site infection | 90 days
  post-operative surgical site infection in patients submitted to Anterior Rectal Resection
Number of participants with abdominal collections | 90 days
  post-operative abdominal collections in patients submitted to Anterior Rectal Resection
Number of participants with anastomotic bleeding | 90 days
  post-operative anastomotic bleeding in patients submitted to Anterior Rectal Resection
Number of participants with perforation | 90 days
  post-operative perforation in patients submitted to Anterior Rectal Resection
Number of participants with anastomotic stenosis | 90 days
  post-operative anastomotic stenosis in patients submitted to Anterior Rectal Resection